CLINICAL TRIAL: NCT03285945
Title: Fluorine-18-fluorodeoxyglucose Uptake in Large-Vessel Giant Cell Arteritis After Short-term, High-Dose Steroid Treatment - A Diagnostic Window of Opportunity?
Brief Title: FDG Uptake in Large-Vessel Giant Cell Arteritis After Short-term, High-Dose Steroid Treatment
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: akutPET
Record Dates: First submitted 2016-10-12; First posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2016-10

CONDITIONS: Giant Cell Arteritis
Keywords: Positron-Emission Tomography
MeSH Terms: conditions — Giant Cell Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Temporal artery biopsies, whole blood, serum, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PET3: Post-therapeutic FDG PET/CT performed after 3 days of steroid treatment
  Interventions: Drug: PET3
- PET10: Post-therapeutic FDG PET/CT performed after 10 days of steroid treatment
  Interventions: Drug: PET10

INTERVENTIONS:
Drug: PET3 — Prednisolone 60 mg daily for 3 days
  Groups: PET3
Drug: PET10 — Prednisolone 60 mg daily for 10 days
  Groups: PET10

SUMMARY:
Giant cell arteritis (GCA) affects large and medium sized vessels. Large vessel-GCA (LV-GCA) affecting aorta and/or its main branches is seen a) together with temporal arteritis (AT-GCA), b) as isolated LV-GCA but also c) with polymyalgia rheumatica.

There is a risk of vision loss and cerebral thromboembolic events or great vessel injury in GCA. With delayed or inadequate treatment mortality and morbidity increases. This highlights the need of fast diagnosis and early treatment.

The cornerstone in the diagnosis of GCA is a positive temporal artery biopsy. Patients with LV-GCA have more general, but less cephalic symptoms than patients with AT-GCA. Also, biopsy from large vessels can rarely be done and only 50% have a positive temporal artery biopsy (TAB). Hence, diagnosis often rely on imaging.

Fluorine-18-fluorodeoxyglucose positron-emission tomography (FDG PET)/CT has shown high diagnostic sensitivity and specificity and is believed to be superior to other imaging modalities in the diagnosis of LV-GCA . The impact of FDG PET/CT in the management of LV-GCA has been evaluated and has shown to increase the diagnostic accuracy in a significant proportion of patients. However, studies have indicated a lower sensitivity in steroid treated patients.

The aim of this study, was to evaluate the effect of steroid treatment on large-vessel FDG uptake in new-onset, treatment-naive LV-GCA by repetitive FDG PET/CT pre- and post therapeutic. With insights into the diagnostic capabilities after treatment is initiated, the possibility of timely treatment and confident diagnostic work up will improve.

DETAILED DESCRIPTION:
As standard of care, patients suspected of GCA undergo clinical examination, laboratory screening, temporal artery biopsy, vascular ultrasound examination and FDG PET/CT.

All patients with a diagnosis of GCA will be treated with 60 mg af prednisolone and tapered according to a predefined algorithm.

In patients with FDG PET/CT verified LV-GCA, FDG PET/CT is repeated after either 3 (n=12) or 10 (n=12) days of steroid treatment.

An experienced nuclear medicine physician (LCG), blinded to clinical symptoms and findings, qualitatively assesses PET scans. A semiquantitative approach is applied (a.m. Meller) in which FDG uptake in vascular regions is graded on a 5-point scale (0 = no uptake, 1 = uptake below or equal to blood pool, 2 = above blood pool but below liver, 3 = above liver, 4 = 2 times above liver). Any score ≥3 is considered consistent with vasculitis. Sensitivity of post-therapeutic FDG PET/CT will be evaluated.

Moreover, standard uptake values (SUV) mean and maximum values in vascular regions will be calculated. A ratio SUV(wall)/SUV(blood pool) and a total metabolic burden (TMB) based on affected vascular volume and SUV mean values are obtained as measures of vascular wall inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical suspicion of GCA; Cranial symptoms, new-onset extremity claudication or protracted constitutional symptoms (weight loss > 5 kilograms or fever >38C for > 3 weeks).
2. C reactive protein >15 mg/l or erythrocyte sedimentation rate >40 mm/h
3. FDG PET/CT verified LV-GCA (steroid-naive) defined by FDG uptake in the aortic wall and/or supra-aortic branches with FDG uptake score ≥3.

Exclusion Criteria:

1. oral glucocorticoid treatment within the past month
2. subcutaneously, intramuscularly, intraarticularly or intravenously administered glucocorticoid within the past 2 months
3. treatment with DMARDs or other immunosuppressive therapy ongoing or within the past 3 months
4. ongoing treatment with interleukin2
5. any disease mimicking GCA, including

   * a) autoimmune diseases with possible aortitis; rheumatoid arthritis, Cogans syndrome, relapsing polychondritis, ankylosing spondylitis, systemic lupus erythematosus, Buerger's disease, Bechet's disease, inflammatory bowel disease
   * b) infections with possible aortitis: syphilis, known active current or history of recurrent tuberculosis, hepatitis or HIV
   * c) other large-vessel disease: sarcoidosis, neurofibromatosis, congenital coarctation, Marfans syndrome, Ehlers-Danlos syndrome, retroperitoneal fibrosis
6. body weight of >150 kg.
7. Previously diagnosed and treated for PMR or GCA

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Steroid-naive, newly-diagnosed giant cell arteritis patients
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2014-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Proportion of large vessel-GCA patients with post-therapeutic FDG uptake consistent with a diagnosis of large vessel giant cell arteritis | Assessed after intervention (3 or 10 days of treatment, respectively)
  Proportion of patients with PET positive large vessel vasculitis defined as vascular FDG uptake≥3, semiquantitative assesment ad modum Meller

SECONDARY OUTCOMES:
Change in quantitive uptake values (SUV) | From baseline to post-treatments scan (3 or 10 days of treatment, respectively)
  The steroid induced change in FDG uptake assessed by; change in maximum standardized uptake values (SUV)
Change in quantitive uptake values (TBR) | From baseline to post-treatments scan (3 or 10 days of treatment, respectively)
  The steroid induced change in FDG uptake assessed by; change in target to background ratio (TBR)= SUVmax(artery)/SUVmean(venous blood pool)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen-Margrethe Hauge, Prof MD PhD, Study Chair — Department of Rheumatology , Aarhus University Hospital
Locations (1):
- Department of Rheumatology, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Puppo C, Massollo M, Paparo F, Camellino D, Piccardo A, Shoushtari Zadeh Naseri M, Villavecchia G, Rollandi GA, Cimmino MA. Giant cell arteritis: a systematic review of the qualitative and semiquantitative methods to assess vasculitis with 18F-fluorodeoxyglucose positron emission tomography. Biomed Res Int. 2014;2014:574248. doi: 10.1155/2014/574248. Epub 2014 Sep 1. PMID 25254211
- [Background] Stellingwerff MD, Brouwer E, Lensen KDF, Rutgers A, Arends S, van der Geest KSM, Glaudemans AWJM, Slart RHJA. Different Scoring Methods of FDG PET/CT in Giant Cell Arteritis: Need for Standardization. Medicine (Baltimore). 2015 Sep;94(37):e1542. doi: 10.1097/MD.0000000000001542. PMID 26376404
- [Background] Fuchs M, Briel M, Daikeler T, Walker UA, Rasch H, Berg S, Ng QK, Raatz H, Jayne D, Kotter I, Blockmans D, Cid MC, Prieto-Gonzalez S, Lamprecht P, Salvarani C, Karageorgaki Z, Watts R, Luqmani R, Muller-Brand J, Tyndall A, Walter MA. The impact of 18F-FDG PET on the management of patients with suspected large vessel vasculitis. Eur J Nucl Med Mol Imaging. 2012 Feb;39(2):344-53. doi: 10.1007/s00259-011-1967-x. Epub 2011 Nov 10. PMID 22072285
- [Background] Prieto-Gonzalez S, Depetris M, Garcia-Martinez A, Espigol-Frigole G, Tavera-Bahillo I, Corbera-Bellata M, Planas-Rigol E, Alba MA, Hernandez-Rodriguez J, Grau JM, Lomena F, Cid MC. Positron emission tomography assessment of large vessel inflammation in patients with newly diagnosed, biopsy-proven giant cell arteritis: a prospective, case-control study. Ann Rheum Dis. 2014 Jul;73(7):1388-92. doi: 10.1136/annrheumdis-2013-204572. Epub 2014 Mar 24. PMID 24665112